CLINICAL TRIAL: NCT02530437
Title: A Phase 1B/2 Study of Taladegib in Combination With Weekly Paclitaxel, Carboplatin, and Radiation in Localized Adenocarcinoma of the Esophagus or Gastroesophageal Junction
Brief Title: Taladegib, Paclitaxel, Carboplatin, and Radiation Therapy in Treating Patients With Localized Esophageal or Gastroesophageal Junction Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor sold the drug TALADEGIB to another company during the trial and thereafter no drug was available. The sponsor made a decision to stop development of this drug Taladegib.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0966; NCI-2015-01554 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0966 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Stage IB Esophageal Adenocarcinoma AJCC v7; Stage II Esophageal Adenocarcinoma AJCC v7; Stage IIA Esophageal Adenocarcinoma AJCC v7; Stage IIB Esophageal Adenocarcinoma AJCC v7; Stage IIIA Esophageal Adenocarcinoma AJCC v7; Stage IIIB Esophageal Adenocarcinoma AJCC v7
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Carboplatin; Radiation; Paclitaxel; Taxes; LY2940680; benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Step I (taladegib, paclitaxel, carboplatin, and radiation) (Experimental): Patients receive taladegib PO for 7 days, followed by taladegib, paclitaxel, carboplatin, and external beam radiation therapy as in Phase IB.
  Interventions: Drug: Carboplatin; Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Taladegib
- Step II (taladegib, paclitaxel, carboplatin, and radiation) (Experimental): Patients receive taladegib, paclitaxel, carboplatin, and external beam radiation therapy as in Phase IB.
  Interventions: Drug: Carboplatin; Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Taladegib

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Taladegib — Given PO
  Other Names: Benzamide, 4-Fluoro-N-methyl-N-(1-(4-(1-methyl-1H-pyrazol-5-yl)-1-phthalazinyl)-4-piperidinyl)-2-(trifluoromethyl)-; LY-2940680; LY2940680

SUMMARY:
This phase IB/II trial studies the side effects of taladegib, paclitaxel, carboplatin, and external beam radiation therapy and to see how well they work in treating patients with esophageal or gastroesophageal junction cancer found only in the tissue or organ where it began, and has not spread to nearby lymph nodes or to other parts of the body (localized). Taladegib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving taladegib, paclitaxel, carboplatin, and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity of taladegib administered orally daily concurrently with weekly paclitaxel, carboplatin and radiation therapy in patients with localized nuclear glioma-associated oncogene homolog (Gli-1) expressing adenocarcinoma of the esophagus or gastroesophageal junction. (Phase IB) II. To assess the rate of pathologic complete response (pathCR) when taladegib is administered orally daily concurrently with weekly paclitaxel, carboplatin, and radiation therapy in patients with localized nuclear Gli-1 expressing adenocarcinoma of the esophagus or gastroesophageal junction. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of biochemoradiation in the phase II study. II. To assess additional biomarkers (hedgehog [Hh] related and Hh unrelated) in sequentially procured tissues (biopsies and resected specimens).

III. Assess if taladegib down modulates its target (Gli-1) in the first cohort (where taladegib will be administered alone for the first 7 days) of the phase II study.

IV. Assess relapse-free survival and overall survival.

OUTLINE:

PHASE IB: Patients receive taladegib orally (PO) once daily (QD) on days 1-38, paclitaxel intravenously (IV) over 3 hours on the first radiation day of each week for 5 doses, carboplatin IV over 2 hours on the first radiation day of each week for 5 doses, and undergo external beam radiation therapy 5 days weekly on 28 consecutive weekdays for 5.5 weeks.

PHASE II: Patients are assigned to 1 of 2 steps.

STEP I: Patients receive taladegib PO for 7 days, followed by taladegib, paclitaxel, carboplatin, and external beam radiation therapy as in Phase IB.

STEP II: Patients receive taladegib, paclitaxel, carboplatin, and external beam radiation therapy as in Phase IB.

After completion of study treatment, patients are followed up at 3 months, every 3-6 months for 1 year, every 6 months for 2 years, and at years 4 and 5.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the esophagus or gastroesophageal junction (EAC)
* Localized EAC and its baseline clinical stage determined as: T2-T3N0 or T1-3N positive (+); imaging studies suspicious for metastases must be followed with a negative biopsy before a patient can enter the study
* Patients with malignant celiac nodes are eligible if the primary lesion is in the mid-thoracic or distal thoracic esophagus or it is involving the gastroesophageal junction
* Tumor must have labeling index of >= 5% of the nuclear Gli-1 (integral biomarker) performed in the MD Anderson Cancer Center Clinical Laboratory Improvement Amendment (CLIA) laboratory for patient to be eligible in this trial (if enough archival tissue is not available to determine labeling index, patient must agree to a biopsy to be eligible for the study)
* Tumor may not extend > 4 cm below the gastroesophageal junction
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* All patients must be willing to provide research tumor tissue for biomarker studies at baseline, from archival tumor tissue or through endoscopy if sufficient archival tissue is not available; all patients must also allow biomarker studies on the tissue obtained through surgery to remove the primary cancer
* Phase II only: patients volunteering for the Phase II part of the protocol must be willing to undergo a research endoscopy for tissue collection on day 8 (+/- 2 days) from the beginning of therapy
* Absolute neutrophil count >= 1500/mm^3
* Platelets greater >= 100,000/mm^3
* Hemoglobin >= 8 g/dL
* Serum creatinine =< 2 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN
* Serum bilirubin =< 1.5 x ULN
* Patient must be able to comprehend the approved consent document and have the willingness to sign it; the patient prior to enrollment and the administration of any protocol-specific therapy must sign the consent document
* Willingness and ability to comply with study procedures and follow-up examinations
* Must be considered medically fit for operation as determined by multidisciplinary evaluation
* Males and females with reproductive potential must agree to use 2 forms of medically approved contraceptive precautions and for at least 6 months following the last dose of biochemoradiation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Women of childbearing potential are defined as follows: having regular menstrual cycles; has amenorrhea, irregular menstrual cycles or using a contraceptive method that precludes withdrawal bleeding; have had a tubal ligation; women are considered not to be of childbearing potential for the following reasons: had hysterectomy and/or bilateral oophorectomy; post-menopausal defined by amenorrhea for at least 1 year in a woman > 45 years old
* Females with childbearing potential must have a negative serum pregnancy test within 14 days prior to treatment start

Exclusion Criteria:

* Baseline clinical stage of T1N0 or inoperable T4 (unequivocal organ involvement) are to be excluded
* Unequivocal metastatic tumor at baseline
* Tracheo-esophageal (TE) fistula or direct invasion into the tracheo-bronchial mucosa; a bronchoscopy (biopsy and cytology should be performed) is required to exclude TE fistula or tracheo-bronchial involvement in patients with a tumor located at < 26 cm from the incisors
* Cervical esophageal cancer will not be entered in this study
* Any prior chemotherapy, surgery, or radiotherapy for EAC
* Prior mediastinal irradiation (for any reason)
* Clinically significant ulcerative colitis, inflammatory bowel disease, or partial or complete small bowel obstruction are to be excluded
* Malabsorption syndrome or other condition that would interfere with intestinal absorption are excluded
* Pregnant or nursing females are to be excluded; breastfeeding should be discontinued if the mother is treated with taladegib
* Presence of other significant cancer(s) or history of other significant cancer(s) within the last 3 years (patients who have been cancer-free for 3 years, or have a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma of the cervix are eligible)
* Known active viral or other chronic types hepatitides (hepatitis B, C) or cirrhosis
* Uncontrolled concurrent illness including, but not limited to: serious uncontrolled infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia that interfere with blood pressure, uncontrolled diabetes, or psychiatric illness/social situations that would limit compliance with the study requirements
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation
* Patients who are receiving concurrent non-protocol anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy, or tumor embolization) are to be excluded
* Patients may not be receiving any other investigational agents
* Patients with known hypersensitivity to taxanes or platinums are to be excluded
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin) are ineligible; patients on strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors will also be excluded
* Known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Any other conditions or circumstances that would, in the opinion of the investigator, make the patient unsuitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer A Ajani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 B: Patient received TALADEGIB PO for 38 days, starting on first chemoradiation day.
Period: Overall Study
Arm/Group | Phase 1 B
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase 1 B
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety of Taladegib When Given in Combination With Paclitaxel, Carboplatin, and Radiation Therapy Defined by Dose-limiting Toxicities (Phase IB)
Description: The safety data will be summarized using frequencies and percentages by adverse event category, grade and attributions.
Time Frame: Up to 5 weeks
Population: Data was not collected
Arm/Group | Phase 1 B
Number analyzed (Participants) | 0

2. Primary Outcome: Pathologic Complete Response Rate (Phase II)
Description: A pathologic complete response (pathCR) rate of at least 35% (>= 40% is desirable) will be of interest. The pathCR rate in each of the treatment step will be estimated, along with the 95% confidence interval.
Time Frame: Up to 4 years and 10 months
Population: 6 had surgery, 1 progressed prior to surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 B
Number analyzed (Participants) | 7
Participants
  Complete Response | 4
  Less than complete response | 3

3. Secondary Outcome: Change in Biomarker Expression Levels of Primary and Secondary Resistance
Description: A linear mixed effect model will be used to assess the change of biomarkers over time. The outcome variable will be biomarker expression level and the covariates will include time, treatment step and time by treatment interaction. The biomarker expression may be log-transformed prior to fit the model in order to satisfy the normality assumption. Also, a logistic regression model will be used for the binary outcome of pathCR, using treatment step, baseline biomarker and the change of biomarker between baseline and at surgery as covariates.
Time Frame: Baseline to the time of surgery
Population: Data was not collected
Arm/Group | Phase 1 B
Number analyzed (Participants) | 0

4. Secondary Outcome: Relapse-free Survival
Description: Kaplan-Meier method will be used to estimate the probabilities of relapse-free survival.
Time Frame: Up to 4 years and 10 months
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1 B
Number analyzed (Participants) | 7
months | 14 [2 to 28]

5. Secondary Outcome: Overall Survival
Description: Kaplan-Meier method will be used to estimate the probabilities of overall survival.
Time Frame: Up to 4 years and 10 months
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1 B
Number analyzed (Participants) | 7
months | 27 [20 to 49]

ADVERSE EVENTS:
Time Frame: Baseline to up to 4 years and 10 months
Groups:
- Phase 1B: Patient received TALADEGIB PO for 38 days, starting on first chemoradiation day.
Arm/Group | Phase 1B
All-Cause Mortality (participants affected / at risk) | 7/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1B (N=7)
Fever (Infections and infestations) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Ischemia cerebrovascular (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1B (N=7)
Nausea (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 2
Lipase increased (Investigations) | 1
Weight loss (Investigations) | 7
Dysgeusia (Nervous system disorders) | 4
Skin changes redness (Skin and subcutaneous tissue disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 6
Dysphagia (Gastrointestinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Right Wrist Pain (Musculoskeletal and connective tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 6
White blood cell decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 5
Chest Pain (Cardiac disorders) | 2
Abdominal cramping (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Hypotension (Vascular disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Visual changes (Eye disorders) | 2
Weakness (General disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Chapped lips (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Mucus (Respiratory, thoracic and mediastinal disorders) | 2
Platelet count decreased (Investigations) | 1
Headache (Nervous system disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Stomach pain (Gastrointestinal disorders) | 1
Flu like symptoms (General disorders) | 1
Fever (General disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Herpes rash (Skin and subcutaneous tissue disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Insomnia (Psychiatric disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal Bloating (Gastrointestinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Post-Nasal Drip (Respiratory, thoracic and mediastinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Anxiety (Psychiatric disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Dysarthria (Nervous system disorders) | 1
Difficulty Coping (Psychiatric disorders) | 1
Palpitations (Cardiac disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Belching (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Right Side Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Right Side Hand Weakness (Nervous system disorders) | 1
Odynophagia (Gastrointestinal disorders) | 5
Pain in extremity (Right Knee) (Musculoskeletal and connective tissue disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic Chest Pain (Cardiac disorders) | 1
Pain in extremity Right Arm (Musculoskeletal and connective tissue disorders) | 1
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1
Skin Dermatitis (Skin and subcutaneous tissue disorders) | 1
Memory impairment (Nervous system disorders) | 1
Ischemia Cerebrovascular (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Taste Alteration: Metallic Taste (Nervous system disorders) | 3
Bruises Easily (Blood and lymphatic system disorders) | 4
Flatulence (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Burping (Gastrointestinal disorders) | 2
Non Cardiac Chest Pain (General disorders) | 1
Substernal Pain (Gastrointestinal disorders) | 1
Hypertension (Vascular disorders) | 1
Light Headedness (Nervous system disorders) | 4
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Burning Chest Pain (Musculoskeletal and connective tissue disorders) | 2
Esophageal Pain (Gastrointestinal disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT02530437/Prot_SAP_000.pdf